CLINICAL TRIAL: NCT07148193
Title: Understanding Long-Term Sarcoma Survivorship: Risk Profiles, Outcomes and Unmet Needs - A Joint Project of Research, Sarcoma Centres and Patient Experts (PROSa+)
Brief Title: Quality of Life and Medical Care of Long-term Sarcoma Survivors in Germany (PROSa+)
Acronym: PROSa+
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Sarcoma Foundation (DSS) (Unknown); German Cancer Research Center (Other); Universitätsmedizin Mannheim (Other); University Hospital, Essen (Other); National Centre for Tumor Diseases Heidelberg (Unknown)
Responsible Party: Principal Investigator, Martin Eichler, Head of the Core Unit Patient-Reported Outcomes at NCT/UCC Dresden, Technische Universität Dresden
Other Study IDs: SR+BO-EK-452112024; 70116152 (Other Grant/Funding Number: Deutsche Krebshilfe)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma; Survivorship; Quality of Life (QOL); Medical Care
Keywords: Sarcoma; Neoplasms; Patient-Reported Outcomes; Patient-Reported Experiences; Medical Care; Quality of Life; Unmet Health Needs; Oncology; Psycho-Oncology
MeSH Terms: conditions — Sarcoma; Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sarcoma survivors: Adults (≥18 years) diagnosed with a sarcoma at least five years prior to study participation, regardless of current disease status, who are treated or receive follow-up care in Germany.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
The study PROSa+ aims to assess patient-reported outcomes (PROs), patient-reported experiences (PREs), and the socioeconomic situation of long-term sarcoma survivors (≥ 5 years post-diagnosis, with or without active disease) in Germany. The mixed-methods research design includes a multicenter observational study with a cross-sectional questionnaire survey involving 1,600 participants (paper, online), qualitative interviews with up to 60 participants, and longitudinal analyses combining data from existing sarcoma registries and the previous PROSa study conducted between 2017 and 2020.

DETAILED DESCRIPTION:
Sarcomas are rare cancers that can arise almost anywhere in the body and account for only about one percent of all cancer diagnoses. Both the disease and its treatments often result in late effects, yet knowledge about these long-term consequences remains limited. The study PROSa+ aims to assess patient-reported outcomes (PROs), patient-reported experiences (PREs), and the socioeconomic situation of long-term sarcoma survivors (≥ 5 years post-diagnosis, with or without active disease) in Germany. Particular focus is placed on subgroups with potential long-term risks, including survivors of bone sarcomas, extremity or trunk sarcomas after multimodal treatment, retroperitoneal sarcomas, gastrointestinal stromal tumors (GIST) with or without long-term TKI therapy, and young adult survivors.

The mixed-methods research design includes a multicenter observational study with a one-time questionnaire survey involving 1,600 participants (paper, online), qualitative interviews with up to 60 participants, and longitudinal analyses combining data from existing sarcoma registries and the previous PROSa study conducted between 2017 and 2020.

Recruitment is built on draws on existing network structures, including the PROSa cohort, the National Center for Tumor Diseases (NCT/UCC) Dresden, the SarcBOP registry at the National Center for Tumor Diseases (NCT) Heidelberg, West German Cancer Center Essen (WTZ), University Hospital Mannheim (UMM), the German Sarcoma Foundation, and cooperating sarcoma centers. Medical data are extracted from patient records.

Statistical analyses will include descriptive statistics and regression models to identify impaired quality of life domains and associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoma according to the International Classification of Diseases for Oncology (ICD-O) and World Health Organization (WHO) classification, including soft tissue sarcoma, bone sarcoma, and GIST
* At least 5 years since initial sarcoma diagnosis
* With or without active disease
* Age ≥18 years at the time of study participation

Exclusion Criteria:

* Diagnosis of Desmoid tumors
* Inability to complete a structured questionnaire (e.g., due to insufficient German language skills, cognitive impairment, dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) diagnosed with a sarcoma at least five years prior to study participation, regardless of current disease status, who are treated or receive follow-up care in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (EORTC QLQ-SURV100) | single-time point (enrollment)
  The EORTC QLQ-SURV100 is a 100-item questionnaire assessing general quality of life among cancer survivors. It includes multiple functional scales covering physical, role, emotional, cognitive, and social functioning, as well as symptom scales (fatigue, pain) and several single-item measures. Most items are rated on a 1-4 scale, while two global items on overall quality of life and general health are rated on a 1-7 scale. Higher scores on the functional and global health status scales indicate better quality of life, whereas higher scores on symptom scales reflect worse quality of life.
  With the exception of five acute symptoms, the SURV100 includes all items from the EORTC QLQ-C30. To enable comparative analyses, the investigators supplemented the SURV100 with these five missing items: appetite loss, nausea, vomiting, constipation, and diarrhea.
Satisfaction with Medical Care (adapted from EORTC OUT-PATSAT7 & self-developed items) | single time point (enrollment)
  Satisfaction with medical care and communication will be assessed using three items adapted from the EORTC OUT-PATSAT7 and three self-developed items, all rated on a 1-5 scale. Higher scores indicate greater satisfaction with the medical care received.
Use of Care Offers (self-developed, adapted from CaSUN) | single time point (enrollment)
  Service utilization will be assessed with self-developed items based on the Cancer Survivors' Unmet Needs measure (CaSUN). Participants indicate their use of 24 different non-rehabilitation care services and 11 rehabilitation care services. Response options include two types of "No" (offer not available or offer available but not used) and, if "Yes," a rating from 1-3 indicating how helpful the offer was, with higher scores reflecting greater helpfulness.
Unmet Needs (self-developed, adapted from CaSUN) | single time point (enrollment)
  Unmet needs will be assessed with self-developed items based on the CaSUN, asking participants about the lack of adequate support or services in 20 areas. Response options include two types of "No" (no need or need has already been met) and, if "Yes," a rating from 1-3 indicating the current intensity of the unmet need, with higher scores reflecting greater unmet need.

SECONDARY OUTCOMES:
Fatigue (EORTC QLQ-FA12) | single-time point (enrollment)
  Fatigue will be assessed using the 12-item EORTC QLQ-FA12 scale, which measures physical, emotional, and cognitive aspects of cancer-related fatigue on a 1-4 scale. Higher scores indicate greater fatigue.
Psychological Distress (PHQ-4) | single-time point (enrollment)
  Psychological distress will be measured using the four-item PHQ-4, including the diagnostic core criteria for depression (PHQ-2) and generalized anxiety disorder (GAD-2), ranging from 1-4. Higher scores indicate greater psychological distress.
Loneliness (UCLA LS-3) | single-time point (enrollment)
  Loneliness will be assessed using the three-item UCLA Loneliness Scale, measuring subjective feelings of loneliness and social isolation, ranging from 1-3. Higher scores indicate greater loneliness.
Physical Complaints (EORTC WISP) | single-time point (enrollment)
  Physical complaints will be measured using the EORTC WISP module, allowing participants to report up to three symptoms and rate the degree of burden from 1-4. Higher scores indicate greater impairment due to the respective symptom.
Communication with Healthcare Professionals (adapted from EORTC COMU26 & self-developed items) | single-time point (enrollment)
  Communication experiences will be assessed using nine items adapted from the EORTC COMU26 and nine self-developed items, focusing on perceived quality and clarity of communication with healthcare providers. Rated on a 1-4 scale, higher scores indicate greater satisfaction with communication.
Information Sources (self-developed, answer options adapted from CaSUN) | single-time point (enrollment)
  Information sources will be assessed using nine self-developed items, asking participants where they obtain cancer-related information. Response options include two types of "No" (not known or known but not used) and, if "Yes," a rating from 1-3 indicating how helpful the source was, with higher scores reflecting greater helpfulness.
Sociodemographic Items | single-time point (enrollment)
  Sociodemographic characteristics, including age, sex, and migration background will be collected.
Socioeconomic Items | single-time point (enrollment)
  Socioeconomic status will be assessed through items measuring i.a. education, employment status, and income.
Physical Activity (adapted Godin-Shephard Leisure-Time Physical Activity Questionnaire) | single-time point (enrollment)
  Physical activity will be measured using an adapted version of the Godin-Shephard Leisure-Time Physical Activity Questionnaire. This 4-item questionnaire evaluates the frequency and duration of mild, moderate and vigorous aerobic activities, as well as moderate-to-vigorous strength training, performed during the week. Scores reflect whether participants meet exercise guidelines:
  * Aerobic guidelines: ≥75 min of vigorous or ≥150 min moderate activity (meeting guidelines) vs. 0-149 minutes of moderatre and vigorous activity per week (not meeting guidelines)
  * Resistance guidelines: ≥2 resistance sessions/week (meeting guidelines) vs. <2 sessions (not meeting guidelines) Higher scores indicate better adherence to physical activity recommendations.
Comorbidities | single-time point (enrollment)
  Information on comorbid conditions (e.g., cardiovascular disease, diabetes, depression) will be collected, capturing co-existing health conditions. The total number of comorbidities will be summed and used as a control variable in the analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Eichler, Dr., Principal Investigator — TU Dresden & NCT/ UCC Dresden; Karen Steindorf, Prof. Dr., Principal Investigator — DKFZ Heidelberg; Richard F. Schlenk, Prof. Dr., Principal Investigator — NCT Heidelberg; Jens Jakob, Prof. Dr., Principal Investigator — Sarcoma Center Mannheim; Uta Dirksen, Prof. Dr., Principal Investigator — University Hospital, Essen; Markus Wartenberg, Principal Investigator — Deutsche Sarkom-Stiftung
Locations (5):
- Germany (5):
  - Technical University Dresden, Dresden, Saxony
  - University Hospital Essen, Essen
  - NCT Heidelberg, Heidelberg
  - Sarcoma Center Mannheim, Mannheim
  - Deutsche Sarkom-Stiftung, Wölfersheim